CLINICAL TRIAL: NCT00567099
Title: Remediation of Schizophrenia Sensory Gating Deficit With Aripiprazole
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: New Mexico VA Healthcare System (U.S. Federal Agency)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Jose M. Canive, MD, New Mexico VA Healthcare System
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0059; BRINM #150
Record Dates: First submitted 2007-12-03; First posted 2007-12-04 (Estimated); Last update posted 2010-05-25 (Estimated); Status verified 2007-12

CONDITIONS: Schizophrenia; Sensory Gating
Keywords: Psychiatry; Antipsychotic; Psychopharmacology; Clinical Trial; Open Label; Schizophrenia; Sensory Gating; Attention; Memory
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Aripiprzole — Dosage form, dosage, frequency and duration:
  Aripiprazole 5-30 mg tabs po qday x 3 months
  Other Names: Aripiprazole (Abilify)

SUMMARY:
The purpose of this study is the use of magnetoencephalography or MEG (a machine that measures magnetic activity in your brain) and electroencephalography or EEG (a technique that measures electrical activity in your brain) to study how sounds are processed in individuals with schizophrenia prior to initiation with aripiprazole treatment and after three months of taking the antipsychotic medication aripiprazole.

DETAILED DESCRIPTION:
Problems with attention and perception are core features of schizophrenia and are hypothesized to result from defects in the filtering or gating of sensory input. Examination of this requires neuroimaging techniques with high temporal resolution. High-density EEG and MEG in combination with structural magnetic resonance imaging (sMRI) are used to map sensory gating. In a number of recent studies patient treated with novel antipsychotics have been shown to have P50 gating ratios resembling those of normal controls rather than that of schizophrenia subjects treatment with conventional antipsychotics. To date, there is no literature on the effects of aripiprzole on sensory gating. Subjects who meet all inclusion criteria will receive a clinical interview, an MRI, MEG, and neuropsychological testing before starting treatment with aripiprazole and again 3 months later to determine if patients with schizophrenia who are treated with aripiprazole will demonstrate a sensory gating ratio similar to normal controls, indicating no deficit in sensory gating

ELIGIBILITY:
Inclusion Criteria:

Patient Population

* Diagnosis of Schizophrenia as determine by the Structured Clinical Interview for DSM-IV
* no comorbid diagnosis of PTSD
* continuous treatment with a conventional antipsychotic, risperidone or olanzapine for at least 3 months
* absence of psychiatric hospitalization for at least 3 month
* no history of drug dependency in their lifetime
* no history of alcohol or other substance abuse in the 6 months prior to entry into the study
* no history of head injury with loss of consciousness for more than 5 minutes
* no history of seizure disorder
* no mood stabilizing agents
* between 18-65 and
* able to sign informed consent

Normal Controls

* Matched in age and gender to patient population
* No history of psychiatric dysfunction or alcohol or other substance dependence in their lifetime as determine by the SCID
* No history of alcohol or other substance abuse in the previous 6 months
* No family history of psychotic disorder in first degree relatives as assessed by the FH-RDC diagnostic interview
* No history of head injury with loss of consciousness for more than 5 minutes
* No history of seizure disorder
* Between 18-65
* Able to sign informed consent

Exclusion Criteria:

Subjects will be excluded from participating in this study if they:

* Require treatment with a mood stabilizer
* Have had an inpatient hospitalization in the past 3 months\
* Have a history of a neurological disorder
* Have any other axis I diagnosis besides schizophrenia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2003-08; Study Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
MEG/EEG and MRI data will be compared with the results of a neuropsych battery and symptom rating scales prior to initiation with aripiprazole and after subject has been on a stable dose of aripiprazole for three month. | MEG/EEG will be repeated after a min. of three months on a stable dose of Aripiprazole

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Canive, MD, Principal Investigator — New Mexico VA Healthcare System / BRINM
Locations (1):
- New Mexico VA Healthcare System, Albuquerque, New Mexico, United States

REFERENCES:
- See also: The New Mexico VA Healthcare System website — http://www.albuquerque.va.gov/
- See also: The website for the Biomedical Research Institute of New Mexico which helps administers the funds for this project — http://www.brinm.org